CLINICAL TRIAL: NCT01248624
Title: Early Specialized Palliative Care Team Intervention for Patients With Metastatic Cancer: A Cluster Randomized Trial
Brief Title: Randomized Controlled Trial of Early Palliative Care for Patients With Advanced Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Cancer Society (CCS) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 06-0525-CE; 17257 and 20509 and 700862 (Other Grant/Funding Number: Canadian Cancer Society)
Record Dates: First submitted 2010-11-22; First posted 2010-11-25 (Estimated); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Cancer
Keywords: Palliative Care; Quality of Life; Satisfaction with Care
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early Palliative Care Referral (Active Comparator): The intervention arm receives early referral to and follow-up by a symptom control and palliative care team at Princess Margaret Hospital.
  Interventions: Behavioral: Early Palliative Care Referral
- Conventional Cancer Care (Placebo Comparator): This control arm receives standard cancer care.
  Interventions: Behavioral: Early Palliative Care Referral

INTERVENTIONS:
Behavioral: Early Palliative Care Referral — The intervention arm receives early referral to and follow-up by a symptom control and palliative care team at Princess Margaret Hospital.

SUMMARY:
Patients with advanced cancer often have numerous physical and psychological symptoms, which can negatively affect their quality of life. A palliative care team of different health care professionals (including doctors, nurses, social workers and therapists) specializes in treating these symptoms and offers support for patients and their families. However, palliative care teams are currently involved only in the last two months of a patient's life or not at all.

The main purpose of this study is to determine whether, compared to conventional cancer care, early involvement by a specialized symptom control and palliative care team in patients with advanced cancer will be associated with: better quality of life, greater patient and caregiver satisfaction with care, better symptom control, improved communication with healthcare providers and improved caregiver quality of life.

DETAILED DESCRIPTION:
Twenty-four cancer outpatient clinics at Princess Margaret Hospital, Toronto have been randomly assigned so that patients attending them will receive either early palliative care (referral to the palliative care team) or routine cancer care.

Patients are recruited from Gastrointestinal, Lung, Genitourinary, Gynecology and Breast clinics and are eligible to participate if they have advanced cancer, and have a life expectancy of six months to two years.

Patients and their caregivers who agree to participate are asked to complete questionnaires at baseline and every month for 4 months. These questionnaires ask about their quality of life, and satisfaction with their medical care. After they have completed the 4-month questionnaires, some patients and their caregivers will be interviewed, so that they can describe in their own words their quality of life, satisfaction with care, and views about palliative care. These interviews will be audiotaped and analyzed to provide additional information that cannot be obtained by questionnaires alone.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Dx of stage IV cancer (metastatic); refractory to hormonal therapy for breast or prostate cancer; stage III or IV for lung cancer.
* ECOG performance status ≤ 2 (estimated by primary oncologist)
* Prognosis of >6 months to 2 years (estimated by primary oncologist)

Exclusion Criteria:

* Insufficient English literacy to complete questionnaires
* Inability of pass the cognitive screening test (SOMC - Short Orientation Memory Concentration test score <20 or >10 errors)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 461 (Actual)
Dates: Start 2006-12; Primary Completion 2011-06 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Patient Heath Related Quality of Life (HRQL) as measured by the FACT-G, QUAL-E and FACIT-Sp. | Three months after enrollment.
  Together, the FACT-G (Functional Assessment of Cancer Therapy-General), QUAL-E (Quality of Life at the End of Life), and FACIT-Sp ('Meaning and Peace' and 'Faith' subscales) measure physical, social/family, emotional, functional and existential well-being.

SECONDARY OUTCOMES:
Symptom control (patient outcome). | Three months after enrollment.
  The patient outcome of 'symptom control' is measured by the ESAS (Edmonton Symptom Assessment System).
Communication with healthcare providers (patient outcome). | 3 months after enrollment.
  Patient communication with healthcare providers is measured by the CARES (Medical Interaction Subscale).
Patient and caregiver satisfaction with care. | 3 months after enrollment.
  The outcome of 'satisfaction with care' is measured by the FAMCARE (Family Satisfaction with Cancer Scale) for primary caregivers. Patients complete a modified version of the FAMCARE scale.
Caregiver quality of life (caregiver outcome). | 3 months after enrollment.
  Caregiver quality of life is measured by Caregiver Quality of Life Index-Cancer (CQOL-C) and the SF-36 (Caregiver Health and Functioning Medical Outcomes Study Short-form).

CONTACTS AND LOCATIONS:
Overall Officials: Camilla Zimmermann, MD, PhD, Principal Investigator — Princess Margaret Cancer Centre, University Health Network
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

REFERENCES:
- [Background] Zimmermann C, Swami N, Krzyzanowska M, Hannon B, Leighl N, Oza A, Moore M, Rydall A, Rodin G, Tannock I, Donner A, Lo C. Early palliative care for patients with advanced cancer: a cluster-randomised controlled trial. Lancet. 2014 May 17;383(9930):1721-30. doi: 10.1016/S0140-6736(13)62416-2. Epub 2014 Feb 19. PMID 24559581
- [Background] McDonald J, Swami N, Hannon B, Lo C, Pope A, Oza A, Leighl N, Krzyzanowska MK, Rodin G, Le LW, Zimmermann C. Impact of early palliative care on caregivers of patients with advanced cancer: cluster randomised trial. Ann Oncol. 2017 Jan 1;28(1):163-168. doi: 10.1093/annonc/mdw438. PMID 27687308
- [Background] Zimmermann C, Swami N, Krzyzanowska M, Leighl N, Rydall A, Rodin G, Tannock I, Hannon B. Perceptions of palliative care among patients with advanced cancer and their caregivers. CMAJ. 2016 Jul 12;188(10):E217-E227. doi: 10.1503/cmaj.151171. Epub 2016 Apr 18. PMID 27091801
- [Derived] Rodin R, Swami N, Pope A, Hui D, Hannon B, Le LW, Zimmermann C. Impact of early palliative care according to baseline symptom severity: Secondary analysis of a cluster-randomized controlled trial in patients with advanced cancer. Cancer Med. 2022 Apr;11(8):1869-1878. doi: 10.1002/cam4.4565. Epub 2022 Feb 9. PMID 35142091
- [Derived] Mah K, Chow B, Swami N, Pope A, Rydall A, Earle C, Krzyzanowska M, Le L, Hales S, Rodin G, Hannon B, Zimmermann C. Early palliative care and quality of dying and death in patients with advanced cancer. BMJ Support Palliat Care. 2023 Oct;13(e1):e74-e77. doi: 10.1136/bmjspcare-2021-002893. Epub 2021 Feb 22. PMID 33619220
- [Derived] Mah K, Swami N, O'Connor B, Hannon B, Rodin G, Zimmermann C. Early palliative intervention: effects on patient care satisfaction in advanced cancer. BMJ Support Palliat Care. 2022 Jun;12(2):218-225. doi: 10.1136/bmjspcare-2020-002710. Epub 2021 Jan 8. PMID 33419858
- [Derived] McDonald J, Swami N, Pope A, Hales S, Nissim R, Rodin G, Hannon B, Zimmermann C. Caregiver quality of life in advanced cancer: Qualitative results from a trial of early palliative care. Palliat Med. 2018 Jan;32(1):69-78. doi: 10.1177/0269216317739806. Epub 2017 Nov 13. PMID 29130418